CLINICAL TRIAL: NCT00482391
Title: Phase II Study of Dose-Dense Doxorubicin and Cyclophosphamide (AC) Followed by Weekly Paclitaxel With Trastuzumab and Lapatinib in HER2/NEU-Overexpressed/Amplified Breast Cancer: Feasibility
Brief Title: Doxorubicin and Cyclophosphamide Followed by Paclitaxel, Trastuzumab, and Lapatinib in Treating Patients With HER2/Neu-Overexpressed Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Dana-Farber Cancer Institute (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-013; MSKCC-07013
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Trastuzumab; Cyclophosphamide; Doxorubicin; Lapatinib; Paclitaxel

ARMS (1):
- AC, PACLITAXEL , TRASTUZUMAB & LAPATINIB (Experimental): The regimen consists of AC (doxorubicin 60 mg/m2, cyclophosphamide 600 mg/m2) q 14 days x 4 with pegfilgrastim, followed by weekly paclitaxel (80 mg/m2) x 12 + trastuzumab (H) + lapatinib (L). Pegfilgrastim 6mg is given subcutaneously (SQ) on day # 2 of each AC. Filgrastim may be used in lieu of pegfilgrastim at the physician's discretion. Trastuzumab will be administered weekly starting with paclitaxel treatment # 1. Near the completion of all chemotherapy, patients may receive trastuzumab on a q 3-weekly schedule, starting as early as with paclitaxel cycle # 12. The total duration of trastuzumab from beginning to end is 52 weeks. Lapatinib will be given orally at 1000 mg daily, starting with trastuzumab for a total duration of 52 weeks. Hormonal therapy such as tamoxifen or an aromatase inhibitor will be given to patients with hormone receptor positive disease at the physician's discretion. Radiation therapy to the breast or chest is recommended to patients as appropriate.
  Interventions: Biological: trastuzumab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: lapatinib ditosylate; Drug: paclitaxel; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: trastuzumab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: lapatinib ditosylate
Drug: paclitaxel
Other: laboratory biomarker analysis

SUMMARY:
The purpose of this study is to study a new treatment for HER-2/neu (+) breast cancer.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Bilateral synchronous breast tumors allowed
  * Any nodal status or tumor size allowed

    * No stage IV disease
* HER2/neu-positive disease

  * 3+ by IHC OR FISH-amplified
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* ECOG performance status 0-1
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.1 mg/dL
* SGOT or SGPT ≤ 2.5 times upper limit of normal (ULN)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and after completion of study therapy
* LVEF ≥ 50% by MUGA scan
* No peripheral neuropathy > grade 1
* No active second malignancy within the past 5 years except for adequately treated nonmelanoma skin cancer or in situ carcinoma of the cervix
* No known allergy or hypersensitivity to doxorubicin hydrochloride, cyclophosphamide, paclitaxel, or other drugs formulated in Cremophor EL
* No psychiatric illness or concurrent medical conditions that would preclude study treatment
* No other conditions, including any of the following:

  * Unstable angina
  * Congestive heart failure
  * Myocardial infarction within the past 12 months
  * High-risk uncontrolled arrhythmias (e.g., ventricular tachycardia, high-grade AV block, or supraventricular arrhythmias that are not adequately controlled)
* No QT prolongation (> 500 ms)
* No active unresolved infections
* No sensitivity to E. coli derived proteins

PRIOR CONCURRENT THERAPY:

* Prior hormonal therapy for chemoprevention allowed
* No prior trastuzumab (Herceptin®)
* No prior anthracyclines
* No concurrent hormonal therapy, including hormonal contraception (e.g., birth control pills or ovarian hormonal or replacement therapy)
* No other concurrent chemotherapy, radiotherapy, immunotherapy, or biotherapy for breast cancer
* No concurrent drugs that may prolong the QT

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2007-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chau T. Dang, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Clifford A. Hudis, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- [Result] Dang C, Lin N, Moy B, Come S, Sugarman S, Morris P, Abbruzzi A, Chen C, Steingart R, Patil S, Norton L, Winer E, Hudis C. Dose-dense doxorubicin and cyclophosphamide followed by weekly paclitaxel with trastuzumab and lapatinib in HER2/neu-overexpressed/amplified breast cancer is not feasible because of excessive diarrhea. J Clin Oncol. 2010 Jun 20;28(18):2982-8. doi: 10.1200/JCO.2009.26.5900. Epub 2010 May 17. PMID 20479410

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AC, PACLITAXEL , TRASTUZUMAB & LAPATINIB
Started | 95
Completed | 92
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | AC, PACLITAXEL , TRASTUZUMAB & LAPATINIB
Number analyzed (Participants) | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 93
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Completed All Planned Therapy
Description: The number of patients who completed all planned therapy (dose-dense adjuvant/ neoadjuvant chemotherapy regimen) in HER-2/neu-overexpressed/ amplified breast cancer patients.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | AC, PACLITAXEL , TRASTUZUMAB & LAPATINIB
Number analyzed (Participants) | 92
participants | 45

2. Secondary Outcome: Number of Patients Who Were Evaluated for Toxicity
Description: Please see adverse event section in the results. Toxicities were assessed by the National Cancer Institute Common Toxicity Criteria (NCI CTC) version 3.0.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-dense Adjuvant/ Neoadjuvant Chemotherapy Regimen
Number analyzed (Participants) | 95
Participants | 95

ADVERSE EVENTS:
Arm/Group | AC, PACLITAXEL , TRASTUZUMAB & LAPATINIB
Serious Adverse Events (participants affected / at risk) | 23/95
Other Adverse Events (participants affected / at risk) | 94/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AC, PACLITAXEL , TRASTUZUMAB & LAPATINIB (N=95)
Cholesterol,high(hypercholestremia) (Metabolism and nutrition disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Edema: limb (Blood and lymphatic system disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Fever (General disorders) | 4 (4)
Flu-like syndrome (General disorders) | 1 (1)
Gastrointestinal, other (Gastrointestinal disorders) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
Inf norm ANC/gr1/2 neut-Cellulitis(skin) (Infections and infestations) | 2 (2)
Inf norm ANC/gr1/2 neut-Gingivitis(oral-gums) (Infections and infestations) | 1 (1)
Inf unknown ANC-Cellulitis(skin) (Infections and infestations) | 1 (1)
Inf unknown ANC-Pneumonia(lung) (Infections and infestations) | 1 (1)
Infection w/ Gr 3/4 neut, Catheter-related (Infections and infestations) | 1 (1)
Infection w/ Gr 3/4 neut, Skin (cellulites) (Infections and infestations) | 1 (1)
Infection, other (Infections and infestations) | 2 (2)
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Liver dysfunction/failure (Hepatobiliary disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Infections and infestations) | 1 (1)
Ocular/Visual - Other (specify) (Eye disorders) | 1 (1)
Pain - Head/headache (General disorders) | 1 (1)
Pain - Muscle (General disorders) | 1 (1)
Pain - Other (specify) (General disorders) | 1 (1)
Pleural effusion (non-malig) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis/pulm infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Prolonged QTc interval (Cardiac disorders) | 1 (1)
Rigors/chills (General disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AC, PACLITAXEL , TRASTUZUMAB & LAPATINIB (N=95)
ALT, SGPT (Metabolism and nutrition disorders) | 22
AST, SGOT (Metabolism and nutrition disorders) | 10
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 6
Constipation (Gastrointestinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 8
Diarrhea (Gastrointestinal disorders) | 50
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6
Fatigue (asthenia, lethargy, malaise) (General disorders) | 49
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 29
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 24
Hemoglobin (Blood and lymphatic system disorders) | 50
Hot flashes/flushes (Endocrine disorders) | 7
Infection (Infections and infestations) | 16
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 9
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 37
Lymphopenia (Blood and lymphatic system disorders) | 38
Mucositis (Clin exam)- Oral cavity (Gastrointestinal disorders) | 12
Nail changes (Skin and subcutaneous tissue disorders) | 7
Nausea (Gastrointestinal disorders) | 18
Neuropathy: sensory (Nervous system disorders) | 16
Neutrophils/granulocytes (ANC/AGC) (Infections and infestations) | 26
Pain - Head/headache (General disorders) | 7
Pain - Other (specify) (General disorders) | 7
Rash/desquamation (Skin and subcutaneous tissue disorders) | 8
Vomiting (Gastrointestinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes